CLINICAL TRIAL: NCT01507792
Title: Effect of Iron Repletion in Women With Chronic Cough and Iron Deficiency
Brief Title: Iron Repletion in Chronic Cough and Iron Deficiency
Acronym: CID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Regione Piemonte (Other)
Responsible Party: Principal Investigator, Caterina Bucca, Associate Professor of Internal Medicine, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRONCOUGH
Record Dates: First submitted 2011-12-29; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Cough; Laryngeal Disease; Bronchial Disease; Iron Deficiency
Keywords: Cough; Laryngismus; Bronchial spasm; Deficiency diseases
MeSH Terms: conditions — Cough; Laryngeal Diseases; Bronchial Diseases; Iron Deficiencies; Laryngismus; Bronchial Spasm; Deficiency Diseases | interventions — Iron-Dextran Complex; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: iron sulphate — 1 or 2 330 mg/daily iron sulphate oral tablets
Drug: antiH1-histamine, proton pump inhibitor — This is not an intervention of interest, but it is a selection criterion to define unexplained cough, as suggested by cough guidelines.
  Other Names: AntiH1-histaminic drug = Loratadine 10 mg; Proton pump inhibitor = omeprazole 20 mg twice daily

SUMMARY:
Chronic cough is more frequent and severe in women than in men. Women often have decreased iron stores, due to menses and pregnancies. Aim of the study: to investigate if iron deficiency has a role in chronic cough by favouring airway hypersensitivity to inhaled irritants.

DETAILED DESCRIPTION:
Women with chronic cough and iron deficiency, cough unresponsive to empiric treatment (suggested by cough guidelines) with antiH1-histaminic drug plus proton pump inhibitor.

Cough VAS (score from 1,best, to 5, worst). Histamine inhalation challenge, performed to assess bronchial, laryngeal, and cough thresholds, performed by delivering doubling concentrations, from 0.5 mg/ml up to 32 mg/ml, by a nebulizer. After each dose FEV1, as bronchial index, maximum mid-inspiratory flow (MIF50) as laryngeal index, and coughs number are assessed. Bronchial threshold is the concentration causing 20% decrease in FEV1, laryngeal threshold that causing 25% decrease in MIF50, cough threshold that causing 5 coughs. Histamine hyperresponsiveness of the bronchi (BHR), larynx (LHR) and cough (coughHR) are defined for thresholds equal or below 8 mg/ml.

Histamine thresholds and cough VAS obtained in baseline, after cough empiric treatment with antiH1-histaminic and proton pump inhibitor, and after iron supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained cough : no detectable trigger for chronic cough identified, such as persistent rhinitis, chronic sinusitis, gastroesophageal reflux disease and asthma.
* no benefit by prior treatment with antiH1-histaminic drug and proton pump inhibitor.
* iron deficiency.
* normal lung function tests and chest radiography no relevant systemic disease.
* no acute respiratory infection in the last eight weeks.
* no pharmacological treatment in the last two weeks.

Exclusion Criteria:

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2002-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change in cough VAS | after 2 months empiric treatment and 2 months iron supplementation
  Changes in cough VAS after 2 months iron supplementation (1 mg/kg elemental iron, corresponding to one or two 330 mg iron sulphate tablets)compared to the value observed after empiric treatment Cough VAS from 0 (best= no cough) to 5 (worst = severe cough)
Change in laryngeal histamine threshold | after 2 months empiric treatment and 2 months iron supplementation
  Change in laryngeal threshold, assessed as the histamine concentration causing 25% decrease from baseline of MIF50 (PC25MIF50), after 2 months iron supplementation (1 mg/kg elemental iron, corresponding to one or two 330 mg iron sulphate tablets), compared to the value obtained after empiric treatment
Change in cough histamine threshold | after 2 months empiric treatment and 2 months iron supplementation
  Change in cough threshold, assessed as the histamine concentration causing 5 or more coughs(PC5cough), after 2 months iron supplementation (1 mg/kg elemental iron, corresponding to one or two 330 mg iron sulphate tablets), compared to the value obtained after empiric treatment

SECONDARY OUTCOMES:
Change in bronchial histamine threshold | after 2 months empiric treatment and 2 months iron supplementation
  Change in bronchial threshold, assessed as the histamine concentration causing 20% decrease from baseline of FEV1 (PC20FEV1), after 2 months iron supplementation (1 mg/kg elemental iron, corresponding to one or two 330 mg iron sulphate tablets), compared to the value obtained after empiric treatment

CONTACTS AND LOCATIONS:
Overall Officials: Caterina B Bucca, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Respiratory Pathophysiology Clinic, ASO San Giovanni Battista, Turin, Italy

REFERENCES:
- [Background] Bucca CB, Bugiani M, Culla B, Guida G, Heffler E, Mietta S, Moretto A, Rolla G, Brussino L. Chronic cough and irritable larynx. J Allergy Clin Immunol. 2011 Feb;127(2):412-9. doi: 10.1016/j.jaci.2010.10.038. Epub 2010 Dec 16. PMID 21167571
- [Background] Bucca CB, Culla B, Guida G, Sciascia S, Bellone G, Moretto A, Heffler E, Bugiani M, Rolla G, Brussino L. Unexplained chronic cough and vitamin B-12 deficiency. Am J Clin Nutr. 2011 Mar;93(3):542-8. doi: 10.3945/ajcn.110.000802. Epub 2011 Jan 19. PMID 21248188
- [Derived] Bucca C, Culla B, Brussino L, Ricciardolo FL, Cicolin A, Heffler E, Bugiani M, Rolla G. Effect of iron supplementation in women with chronic cough and iron deficiency. Int J Clin Pract. 2012 Nov;66(11):1095-100. doi: 10.1111/ijcp.12001. PMID 23067033